CLINICAL TRIAL: NCT01748968
Title: Veterans Living With HIV/AIDS: A Pilot Study Examining Risk Factors Associated With Self-Directed Violence
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: Public Health Grant Program, Veterans Health Administration Office of Public Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-0755
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2012-12

CONDITIONS: Human Immunodeficiency Virus Infection(HIV)/Acquired Immunodeficiency Syndrome (AIDS); Self-Directed Violence
Keywords: Veterans; Human Immunodeficiency Virus Infection(HIV)/Acquired Immunodeficiency Syndrome (AIDS); Self-Directed Violence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Veterans with HIV/AIDS: Veterans with HIV/AIDS

SUMMARY:
The purpose of this project is to gather pilot data related to risk factors associated with suicide in Veterans with Human Immunodeficiency Virus (HIV)/ Acquired Immune Deficiency Syndrome (AIDS) and to develop an educational and interventional tool and instructional guide that can be utilized by local and national providers to increase understanding regarding suicide risk assessment. There are no hypotheses associated with this qualitative pilot study.

DETAILED DESCRIPTION:
To achieve these goals, a semi-structured interview will be conducted to gather this qualitative information. Specifically, this study aims to gather the following information from Veterans with HIV/AIDS: a) information regarding disease acquisition; b) psychosocial stressors; c) social supports; d) protective factors; and e) previous suicidal ideation and behaviors. Further, additional exploratory questions will be asked regarding proposed modifications to the Suicide Risk Assessment Guide Pocket Card, an existing VA tool, so that it can be modified for use by local and national HIV/AIDS providers.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 to 90
* Have a diagnosis of HIV/AIDS
* Currently receiving HIV/AIDS treatment
* Currently receiving or eligible to receive physical and/or mental health care through the VA Eastern Colorado Health Care System

Exclusion Criteria:

* Psychosis at time of interview as determined by observation and/or interview.
* Intoxication via alcohol or other illicit drugs at time of assessment as determined by observation and/or interview.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans with HIV/AIDS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Interview | Interview conducted one time per participant (completion time: approximately 1 hour)
  Semi-structured interview will be utilized to gather the following information from Veterans with HIV/AIDS: a) information regarding disease acquisition; b) psychosocial stressors; c) social supports; d) protective factors; and e) previous suicidal ideation and behaviors. Further, additional exploratory questions will be asked regarding proposed modifications to the Suicide Risk Assessment Guide Pocket Card, an existing VA tool, so that it can be modified for use by local and national HIV/AIDS providers.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Signoracci, Ph.D., Principal Investigator — VISN 19 Denver VA MIRECC
Locations (1):
- Denver VA, Denver, Colorado, United States